CLINICAL TRIAL: NCT03289481
Title: Treatment of HFpEF With Nitrate Supplement: A Double-blind, Placebo Controlled Trial Including Patients With Atrial Fibrillation
Brief Title: Treatment of HFpEF With Nitrate Supplement
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: MaineHealth (Other)
Collaborators: HumanN (Industry)
Responsible Party: Principal Investigator, Ralph Hamill, Cardiologist, MaineHealth
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Neo40 Study
Record Dates: First submitted 2017-09-18; First posted 2017-09-21 (Actual); Results first posted 2019-08-26 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Heart Failure With Normal Ejection Fraction
Keywords: Heart failure; HFpEF; Nitrate supplement
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo controlled crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking will be done by the pharmacy. Active and placebo lozenges will look identical.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active lozenge first (Active Comparator): Subject will take active lozenge (Vitamin C, Vitamin B12, Nitric Oxide Blend, L-citrulline, Sodium Nitrite) for one week, perform cardiac testing then take placebo lozenge for one week and perform cardiac testing.
  Interventions: Dietary Supplement: Active lozenge; Drug: Placebo
- Placebo lozenge first (Active Comparator): Subject will take placebo lozenge for one week, perform cardiac testing then take active lozenge (Vitamin C, Vitamin B12, Nitric Oxide Blend, L-citrulline, Sodium Nitrite) for one week and perform cardiac testing.
  Interventions: Dietary Supplement: Active lozenge; Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Active lozenge — nitric oxide generating lozenge
Drug: Placebo — placebo tablet

SUMMARY:
The objective of this project is to determine if Neo40, a nitric oxide generating lozenge, when consumed twice daily by subjects with HFpEF, will increase exercise tolerance, decrease symptoms and improve quality of life for patients.

DETAILED DESCRIPTION:
Heart failure (HF) is the most common principal diagnosis for hospital admission in patients over 65 years old. There are two types of HF, those with reduced ejection fraction (HFrEF) and those with preserved ejection fraction (HFpEF). Approximately half of patients with the clinical syndrome of HF have preserved systolic function. HEpEF is becoming more prevalent with aging of the population and obesity. There are only two class I recommendations for the treatment of HFpEF, which are controlling blood pressure and the use of diuretics to relieve symptoms. Exercise training is another approach to improving symptoms, however it may be poorly tolerated.

Nitrate supplement in the form of concentrated beetroot juice was recently shown to improve exercise tolerance in patients with HFpEF. (1) Beetroot juice contains high concentration of nitrate (NO3). This is metabolized to nitrite (NO2). It enters the blood stream, where it is further reduced to nitric oxide (NO) resulting in intense vasodilation.

Patients with diastolic dysfunction are often asymptomatic at rest but complain of dyspnea with exertion. Increase in heart rate with exercise causes reduced diastolic filling time and increases left sided filling pressure. Borloug, et al demonstrated this with right heart catheterization and supine exercise in patients with diastolic dysfunction. Infusion of NO2 resulted in decreased filling pressures and increased cardiac output. (2)

Neo40 is a new product made from concentrated beetroot juice in the form of a lozenge designed to dissolve on the tongue. NO3 supplement causes vasodilatation only in the setting of hypoxia and acidosis resulting in targeted vasodilatation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HFpEF, defined as:

   * symptomatic with one of more of the following: orthopnea, paroxysmal nocturnal dyspnea, lower-extremity edema, dyspnea on exertion; AND
   * ejection fraction >50%
   * ratio of early mitral inflow velocity to septal tissue dopler velocity >8; AND
   * one or more of the following: left atrium measurement >34 mL/m2, elevated N-terminal pro-brain natriuretic peptide level within the past 12 months, long term loop diuretic use for control of symptoms or elevated filling pressures on prior cardiac catheterization
2. Stable medical therapy, defined as: no change in cardiac medications within 30 days
3. Willing to comply with the protocol and provide written informed consent

Exclusion Criteria:

1. Non-cardiac condition causing limitation of exercise tolerance
2. Acute coronary syndrome, myocardial infarction or cardiac revascularization within 60 days
3. Clinically significant valvular disease, defined as moderate-severe or severe stenosis or insufficiency
4. Significant ischemia seen on stress testing within the past 12 months that was not revascularized
5. Subject has taken and investigational medication within the past 30 days
6. History of allergy to beets
7. Systolic blood pressure of <100 at screening
8. Significant medical condition that would interfere with treatment, safety or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Hamill, MD, Principal Investigator — MaineHealth
Locations (1):
- Penobscot Bay Medical Center, Rockport, Maine, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eggebeen J, Kim-Shapiro DB, Haykowsky M, Morgan TM, Basu S, Brubaker P, Rejeski J, Kitzman DW. One Week of Daily Dosing With Beetroot Juice Improves Submaximal Endurance and Blood Pressure in Older Patients With Heart Failure and Preserved Ejection Fraction. JACC Heart Fail. 2016 Jun;4(6):428-37. doi: 10.1016/j.jchf.2015.12.013. Epub 2016 Feb 10. PMID 26874390
- [Background] Borlaug BA, Koepp KE, Melenovsky V. Sodium Nitrite Improves Exercise Hemodynamics and Ventricular Performance in Heart Failure With Preserved Ejection Fraction. J Am Coll Cardiol. 2015 Oct 13;66(15):1672-82. doi: 10.1016/j.jacc.2015.07.067. PMID 26449137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a cross over case-control study (each subject was a control for themselves).
Groups:
- Active Lozenge First: Subject will take active lozenge for one week, perform cardiac testing then take placebo lozenge for one week and perform cardiac testing.
  Active lozenge: nitric oxide generating lozenge
- Placebo Lozenge First: Subject will take placebo lozenge for one week, perform cardiac testing then take active lozenge for one week and perform cardiac testing.
  Active lozenge: nitric oxide generating lozenge
Period: Overall Study
Arm/Group | Active Lozenge First | Placebo Lozenge First
Started | 6 | 7
Completed | 4 | 5
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Lozenge First | Placebo Lozenge First | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9
Diagnosis of HFpEF [Count of Participants; unit: Participants] | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Time on Treadmill
Description: change in total time traveled on treadmill
Time Frame: after one week of active lozenges compared to one week of placebo lozenges
Measure: Mean (Full Range); unit: seconds
Groups:
- Active Lozenge: Participants who received Neo40 (active lozenge) in either the first week or the last week of the study.
- Placebo: Participants who received the placebo (matching Neo40) in either the first week or the last week of the study.
Arm/Group | Active Lozenge | Placebo
Number analyzed (Participants) | 9 | 9
seconds | 402.8 [156 to 729] | 181.2 [180 to 660]

2. Primary Outcome: Metabolic Equivalents
Description: change in metabolic equivalents on treadmill
Time Frame: after one week of active lozenges compared to one week of placebo lozenges
Measure: Mean (Full Range); unit: cal/min
Arm/Group | Active Lozenge | Placebo
Number analyzed (Participants) | 9 | 9
cal/min | 7.99 [4.2 to 12.8] | 8.46 [4.2 to 12.8]

3. Primary Outcome: E/E Prime
Description: change in E/E prime on exercise echo (E/E prime is a ratio between early mitral inflow velocity and mitral annular early diastolic velocity in order to measure diastolic dysfunction)
Time Frame: after one week of active lozenges compared to one week of placebo lozenges
Measure: Mean (Full Range); unit: ratio
Groups:
- Placebo Lozenge: Participants who received the placebo (matching Neo40) in either the first week or the last week of the study.
Arm/Group | Active Lozenge | Placebo Lozenge
Number analyzed (Participants) | 9 | 9
ratio | 1.93 [-6.2 to 8] | -.05 [-6.8 to 2.4]

4. Primary Outcome: Estimated Right Ventricular Systolic Pressure
Description: change in estimated right ventricular systolic pressure on echo
Time Frame: after one week of active lozenges compared to one week of placebo lozenges
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Active Lozenge | Placebo
Number analyzed (Participants) | 9 | 9
mmHg | 11.79 [5 to 27] | 8.6 [-1.2 to 28]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Active Lozenge | Placebo Lozenge
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

LIMITATIONS AND CAVEATS:
Low enrollment number

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT03289481/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT03289481/SAP_001.pdf